CLINICAL TRIAL: NCT01724983
Title: Effects of Ketamine on Recovery From Bariatric Surgery
Brief Title: Ketamine in Bariatric Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KET2271
Record Dates: First submitted 2012-09-14; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Morbid Obesity
Keywords: pain; mood; depression; respiration
MeSH Terms: conditions — Obesity, Morbid; Pain; Depression; Respiratory Aspiration | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine (Experimental): patients will receive ketamine at induction
  Interventions: Drug: ketamine
- fentanyl (Active Comparator): patients will receive fentanyl at induction
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: ketamine
  Arms: ketamine
Drug: fentanyl
  Arms: fentanyl

SUMMARY:
Ketamine may improve recovery from bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* obesity (Body Mass Index > 30)
* ASA classificazion < 4
* candidate to bariatric surgery

Exclusion Criteria:

* known or presumed pregnancy
* previous surgery on the airway, esophagus or stomach
* uncontrolled psychiatric symptomatology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
pain level | postoperatively, up to 3 months
mood level | postoperatively, up to 3 months

SECONDARY OUTCOMES:
total dosages of analgesic and muscle relaxant drugs | postoperatively, up to 3 months
postanesthetic recovery | postoperatively, up to 24 hours
satisfaction of the patient and of the surgeon | day 1
pulse oximetry saturation | postoperatively, up to 24 hours
lung volumes | postoperatively, up to 48 hours from end of surgery
antihemetic drug dosage | postoperatively, up to 24 hours
vasoactive drugs | intraoperatively and up to 24 hours from surgery end

CONTACTS AND LOCATIONS:
Overall Officials: Ulderico Freo, MD, Principal Investigator — University of Padova
Locations (1):
- Azienda Ospedaliera, Padua, PD, Italy